CLINICAL TRIAL: NCT06264297
Title: High-Voltage Pulsed Radiofrequency of the Lumbar Dorsal Root Ganglion for the Treatment of Chronic Lumbar Radicular and Neuropathic Pain; A Prospective, Doble-blinded and Randomized Controlled Trial
Acronym: Radiofrequency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Maria Martinez, Anesthesiologist, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01-22-270-111
Record Dates: First submitted 2024-02-12; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Pulsed Radiofrequency; Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I (Active Comparator): RFP on the affected level or levels will be carried out during three cycles of 120 s, limited to a temperature of 42° and a voltage of 45V
  Interventions: Procedure: Radiofrequency
- GROUP II (Experimental): RFP on the affected level or levels will be carried out during three cycles of 120 s, limited to a temperature of 42° and a voltage of 65V
  Interventions: Procedure: Radiofrequency

INTERVENTIONS:
Procedure: Radiofrequency — Pulsed radiofrequency (PRF) is a nonablative pain treatment that uses radiofrequency current in short high-voltage bursts, resulting in interruption of nociceptive afferent pathways. This study aims to show how the variation in radiofrequency voltage applied to the dorsal root ganglion (DRG) affects the treatment of neuropathic pain.

SUMMARY:
The management of chronic lumbar radicular and neuropathic pain is complex and the treatment success rates are low. Pulsed radiofrequency (PRF) has been described in these cases. In order to determine whether high-voltage PRF show better results than PRF a prospective, doble-blinded and randomized study is conducted in patients with chronic lumbar radicular and neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Unilateral pain radiating to the lower extremity (with or without lumbar pain), which clinically corresponds to the path of the corresponding dermatomes.
* Correlation between clinical symptoms and lesion observed by magnetic resonance imaging (MRI).
* Radicular syndrome of three months or more of evolution.
* Normal or pathological electromyogram (EMG).
* Pain with neuropathic characteristics confirmed by the DN4 neuropathic pain questionnaire.
* Patients with a previous positive block diagnosis.
* Patients who have signed the informed consent document.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with non-radicular low back pain.
* MRI not consistent with the patient's symptoms.
* Patients with peripheral neuropathy of the lower extremities.
* Patients with a history or current diagnosis of serious mental disorder.
* Patients with moderate or severe cognitive impairment, or evidence of acute or subacute confusional syndrome.
* Infection at the puncture site.
* Coagulation disorders.
* Pregnant patients.
* Patients who refuse to sign the informed consent document.
* Patients allergic to radiological contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
OSWESTRY LOW BACK DISABILITY QUESTIONNAIRE | From enrollment to the end of treatment at 6 months
  this questionnaire has been designed to give us information as to how your back pain has affected your ability to manage everyday life

SECONDARY OUTCOMES:
DN4 - QUESTIONNAIRE | From enrollment to the end of treatment at 6 months
  DN4 - QUESTIONNAIRE To estimate the probability of neuropathic pain, please answer yes or no for each item of the following four questions.
Visual Numeric Scale | From enrollment to the end of treatment at 6 months
  ranging from 0 to 10 was used to measure pain intensity
Categorical scale | From enrollment to the end of treatment at 6 months
  uses adjectives, such as "mild," "moderate," "severe," and excruciating," to describe pain levels.
patient global impression of improvement (pgi-i) score | From enrollment to the end of treatment at 6 months
  is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erdine S, Bilir A, Cosman ER, Cosman ER Jr. Ultrastructural changes in axons following exposure to pulsed radiofrequency fields. Pain Pract. 2009 Nov-Dec;9(6):407-17. doi: 10.1111/j.1533-2500.2009.00317.x. Epub 2009 Sep 15. PMID 19761513
- [Background] Ewertowska E, Mercadal B, Munoz V, Ivorra A, Trujillo M, Berjano E. Effect of applied voltage, duration and repetition frequency of RF pulses for pain relief on temperature spikes and electrical field: a computer modelling study. Int J Hyperthermia. 2018 Feb;34(1):112-121. doi: 10.1080/02656736.2017.1323122. Epub 2017 May 16. PMID 28540817
- [Background] Cosman ER Jr, Cosman ER Sr. Electric and thermal field effects in tissue around radiofrequency electrodes. Pain Med. 2005 Nov-Dec;6(6):405-24. doi: 10.1111/j.1526-4637.2005.00076.x. PMID 16336478
- [Background] Russo M, Santarelli D, Wright R, Gilligan C. A History of the Development of Radiofrequency Neurotomy. J Pain Res. 2021 Dec 24;14:3897-3907. doi: 10.2147/JPR.S334862. eCollection 2021. PMID 34992451
- [Background] Abejon D, Garcia-del-Valle S, Fuentes ML, Gomez-Arnau JI, Reig E, van Zundert J. Pulsed radiofrequency in lumbar radicular pain: clinical effects in various etiological groups. Pain Pract. 2007 Mar;7(1):21-6. doi: 10.1111/j.1533-2500.2007.00105.x. PMID 17305674
- [Background] Van Boxem K, Huntoon M, Van Zundert J, Patijn J, van Kleef M, Joosten EA. Pulsed radiofrequency: a review of the basic science as applied to the pathophysiology of radicular pain: a call for clinical translation. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):149-59. doi: 10.1097/AAP.0000000000000063. PMID 24553305
- [Background] Vigneri S, Sindaco G, La Grua M, Zanella M, Lo Bianco G, Paci V, Vinci FM, Sciacca C, Ravaioli L, Pari G. Electrocatheter-mediated High-voltage Pulsed Radiofrequency of the Dorsal Root Ganglion in the Treatment of Chronic Lumbosacral Neuropathic Pain: A Randomized Controlled Study. Clin J Pain. 2020 Jan;36(1):25-33. doi: 10.1097/AJP.0000000000000766. PMID 31577546
- [Background] Van Boxem K, van Bilsen J, de Meij N, Herrler A, Kessels F, Van Zundert J, van Kleef M. Pulsed radiofrequency treatment adjacent to the lumbar dorsal root ganglion for the management of lumbosacral radicular syndrome: a clinical audit. Pain Med. 2011 Sep;12(9):1322-30. doi: 10.1111/j.1526-4637.2011.01202.x. Epub 2011 Aug 3. PMID 21812907
- [Background] Karakose Caliskan D, Akesen S, Turker YG, Gurbet A. The effect of combined pulsed radiofrequency treatment to dorsal root ganglion with transforaminal epidural steroid injection on pain. Agri. 2021 Oct;33(4):223-231. doi: 10.14744/agri.2021.94824. PMID 34671961
- [Background] Vuka I, Marcius T, Dosenovic S, Ferhatovic Hamzic L, Vucic K, Sapunar D, Puljak L. Efficacy and Safety of Pulsed Radiofrequency as a Method of Dorsal Root Ganglia Stimulation in Patients with Neuropathic Pain: A Systematic Review. Pain Med. 2020 Dec 25;21(12):3320-3343. doi: 10.1093/pm/pnaa141. PMID 32488240
- [Background] De M, Mohan VK, Bhoi D, Talawar P, Kumar A, Garg B, Trikha A, Dehran M, Kashyap L, Shende DR. Transforaminal Epidural Injection of Local Anesthetic and Dorsal Root Ganglion Pulsed Radiofrequency Treatment in Lumbar Radicular Pain: A Randomized, Triple-Blind, Active-Control Trial. Pain Pract. 2020 Feb;20(2):154-167. doi: 10.1111/papr.12840. Epub 2019 Oct 21. PMID 31538405
- [Background] Napoli A, Alfieri G, Scipione R, Andrani F, Leonardi A, Catalano C. Pulsed radiofrequency for low-back pain and sciatica. Expert Rev Med Devices. 2020 Feb;17(2):83-86. doi: 10.1080/17434440.2020.1719828. Epub 2020 Jan 23. No abstract available. PMID 31973587